CLINICAL TRIAL: NCT07319728
Title: Novel Transdermal Ketoprofen Gel Formulation for Knee Osteoarthritis: Comprehensive In-Vitro and Clinical Assessment
Brief Title: Novel Transdermal Ketoprofen Gel Formulation for Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Hamed Mohie Eldin, Associate professor Clinical pharmacy department, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Minia University
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee joint osteoarthritis; Transdermal Ketoprofen Gel
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- formulation arm (Experimental): new formulation of ketoprofen
  Interventions: Drug: ketoprofen
- commercial product (Active Comparator): positive control receiving commercial product
  Interventions: Drug: ketoprofen

INTERVENTIONS:
Drug: ketoprofen — new gel formulation
  Arms: formulation arm
Drug: ketoprofen — commercial gel
  Arms: commercial product

SUMMARY:
A single blind randomized controlled clinical study

DETAILED DESCRIPTION:
A single blind randomized controlled clinical study

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with osteoarthritis in knee by:

Full history taking Physical examination including (joint tenderness, swelling, crepitus and limitation of motion).

Exclusion Criteria:

* 1. Patients with dual diagnosis 2. Patients have skin lesion or dermatologic disease in the treatment area

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-05-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 weeks
McMaster Universities Arthritis Index (WOMAC) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Hassan, Principal Investigator — Badr University
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Fan M, Wang H, You Y, Wei C, Liu M, Luo A, Xu X, Duan X. Relative safety and efficacy of topical and oral NSAIDs in the treatment of osteoarthritis: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Sep 9;101(36):e30354. doi: 10.1097/MD.0000000000030354. PMID 36086745